CLINICAL TRIAL: NCT05881642
Title: Robot-assisted Cystectomy With Prostate and Seminal-sparing Technique Followed by Modified Orthotopic Ileal Neobladder
Brief Title: Robot-assisted Function-sparing Cystectomy Followed by Modified Orthotopic Ileal Neobladder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0857-01
Record Dates: First submitted 2023-04-25; First posted 2023-05-31 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Negative Surgical Margins
MeSH Terms: conditions — Margins of Excision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate and seminal-sparing Cystectomy (Experimental): Patients undergoing transurethral resection and enucleation of the prostate before robot-assisted cystectomy
  Interventions: Procedure: Prostate and seminal-sparing Cystectomy
- Conventional Radical Cystoprostatectomy (Placebo Comparator): Patients undergoing conventional robot-assisted radical cystoprostatectomy
  Interventions: Procedure: Conventional Radical Cystoprostatectomy

INTERVENTIONS:
Procedure: Prostate and seminal-sparing Cystectomy — Adopt endoscopic enucleation technology to preserve the prostate capsule and part of the urinary control support structure to help restore urinary control and erectile functions
  Arms: Prostate and seminal-sparing Cystectomy
Procedure: Conventional Radical Cystoprostatectomy — According to the consensus standard program, remove the accessory tissues including the bladder,prostate and seminal vesicles
  Arms: Conventional Radical Cystoprostatectomy

SUMMARY:
With the same tumor control rate as classic radical cystectomy, radical cystectomy with partial preservation of the prostate and seminal vesicle can effectively preserve penile erection and fertility, improve urinary control rate and shorten hospitalization time. In this project, transurethral resection of the prostate was used to remove part of the prostate, which further reduced the trauma of radical cystectomy and better preserved the nerves and urethral sphincter. Rapid intraoperative examination of resected tissue can provide a basis for the selection of surgical options. Robot-assisted radical cystectomy can perform pelvic lymph node dissection more accurately, preserve neurovascular complex more effectively, and improve the control effect of tumor and the protective effect of sexual function and reproductive function. In view of the shortcomings of the internationally accepted orthotopic ileal neobladder, this study improved the operation according to the physiological and anatomical characteristics, restored the orthophoria of the new bladder, maintained the consistency of physiological anatomy, and minimized the bladder pressure.

DETAILED DESCRIPTION:
Interventional group：patients undergoing transurethral resection and enucleation of the prostate first, do not open the bladder neck to maintain the integrity of the bladder neck. The enucleated prostate capsule and seminal vesicle are preserved under robotic surgery, and the urinary catheter is stretched during the operation to avoid implantation and metastasis.

Conventional group：patients undergoing conventional robotic radical cystoprostatectomy. All the patients undergoing cystectomy and accept at least 12 months follow up.

Followup: Each patient was evaluated at 3-month intervals for 1 year, at 6- month intervals for 2 to 3 years. Renal ultrasound, biochemical examination and urine culture were done every 3 to 6 months. Pelvic computerized tomography and retro-cystogram were performed 6 months postoperatively and annually thereafter. Urodynamic investigation and cystoscopic examination were done annually.

Postoperative complications were classified as early (90 days or less) and late (greater than 90 days). Early and late complications were subdivided into those related and not related to the neobladder. Major complications were defined as grade III or higher.

Daytime and nighttime continence levels were recorded postoperatively at patient interview. Continence was defined as complete if the patient was dry without a pad, satisfactory if no more than 1 pad was required and poor if the patient used more than 1 pad during the day or night.

ELIGIBILITY:
Inclusion Criteria:

1. Muscle invasive or recurrent multiple non-muscle invasive bladder cancer patients
2. Invasive bladder cancer patients without invasion of the triangle and posterior urethra
3. Age < 70 years old, urethral sphincter function is good
4. Male patients with serum prostate specific antigen < 4ug / L

Exclusion Criteria:

1. Possible recurrence of urethra after cystectomy
2. Patients with bladder adenocarcinoma and squamous cell carcinoma should not undergo orthotopic neobladder.
3. Patients with renal insufficiency
4. Severe liver dysfunction
5. Severe intestinal diseases ( Crohn 's disease, short bowel syndrome )
6. Preoperative tumor breaks through the bladder and invades the surrounding tissue
7. urethral stricture cannot pass through the resectoscope

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only male patient have prostate
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative urinary function | During each follow-up postoperatively, the assessment is evaluated 36 months postoperatively
  Assess post-operative urinary function

SECONDARY OUTCOMES:
bladder cancer specific survival rate | During each follow-up postoperatively, the assessment is calculated based on the 36 months result postoperatively
  Determine bladder cancer control as measured by margin status and time to disease recurrence
Sexual function | During each follow-up postoperatively, the assessment is calculated based on the BCI score of 36 months postoperatively
  Assess post-operative sexual function

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Zhang, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union hospital,Tongji medical college, Huazhong university of science and techonology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No